CLINICAL TRIAL: NCT01310972
Title: Adjuvant Colon Cancer With ELOXatin®/5 FU Based Regimen: ACCELOX
Brief Title: Adjuvant Colon Cancer w/ ELOXatin®/5 FU Based Regimen: ACCELOX
Status: Completed | Type: Observational
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: RAC# 2071-027; RAC# 2071-027 (Other: KFSH&RC IRB)
Record Dates: First submitted 2011-03-06; First posted 2011-03-09 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Colon Cancer
Keywords: Adjuvant Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Registry — Registry

SUMMARY:
Adjuvant Colon Cancer With ELOXatin®/5 FU Based Regimen: ACCELOX

DETAILED DESCRIPTION:
It's a study of adjuvant colon carcinoma using ELOXatin/5-FU based chemotherapeutic regimen called ACCELOX as a definitive curative therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Adjuvant Colon Cancer

Exclusion Criteria:

* Patients with diagnosis other than Colon Cancer.

Ages: 14 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Colon Cancer Registry
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2007-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
OS, PFS, DFS | For the duration of the experiment

CONTACTS AND LOCATIONS:
Overall Officials: Al Jubran, M.D., Principal Investigator — KFSH & RC
Locations (1):
- Kfsh & Rc, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided